CLINICAL TRIAL: NCT00083512
Title: Urinary and Serum VEGF and MMP Levels in Patients Receiving Radiation Therapy for Glioblastoma Multiforme: Prospective Determination of a Predictive Value for Recurrence
Brief Title: Collection of Blood and Urine Samples in Patients Receiving Radiation Therapy for Glioblastoma Multiforme
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040200; 04-C-0200; NCT00087308 (obsolete NCT alias)
Record Dates: First submitted 2004-05-25; First posted 2004-05-25 (Estimated); Last update posted 2025-12-31 (Actual); Status verified 2025-12-16

CONDITIONS: Glioblastoma Multiforme
Keywords: Blood; Urine; GBM; Radiation; Natural History; Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/Glioblastoma multiforme patients: Patients with histologically confirmed supratentorial Glioblastoma multiforme

SUMMARY:
This study will collect blood and urine samples from patients undergoing radiation therapy for glioblastoma multiforme (a type of brain tumor) to investigate the effects of this treatment on blood cells and certain proteins. The information from this study may help scientists develop new tests to measure radiation exposure and find new ways to treat cancer with radiation, and help determine which kinds of patients or tumors respond better to radiation therapy. Two proteins of particular interest in this study and which may be involved in the recurrence of cancer are VEGF (vascular endothelial growth factor) and MMPs (matrix metalloproteinases).

Patients 18 years of age and older with glioblastoma multiforme who are receiving or will receive radiation therapy as part of their medical treatment may be eligible for this study. Candidates are screened with a history and physical examination, blood tests, and magnetic resonance imaging (MRI) of the brain.

Participants will have blood and urine samples collected before, during and after completion of their radiation treatment. Urine samples are collected in a cup and about 2 tablespoons of blood are withdrawn through a needle in a vein. Additional samples may be requested at different times during treatment and in the 3-year follow-up period.

DETAILED DESCRIPTION:
BACKGROUND

* Preliminary data generated from our pilot protocol 02-C-0064 suggests that the urinary VEGF and MMP level at the one month follow-up time point compared to the last on-treatment time point collection may be predictive of tumor recurrence at one year.
* Note that this preliminary study included patients with all histologies.
* In an ongoing effort to validate our results with a larger more homogeneous patient cohort we propose to prospectively study patients undergoing radiotherapy for GBM.

OBJECTIVES

-We will determine whether VEGF and MMP level measurements aid in predicting tumor recurrence at 1 year.

ELIGIBILITY

-Patients seen in the radiation oncology clinic will be asked to provide samples of blood and urine before, during and after their radiation treatment.

DESIGN

* This protocol-provides a means of acquiring blood and urine samples from patients receiving radiation therapy for Glioblastoma multiforme (GBM).
* Patients will be analyzed according to their Radiation Therapy Oncology Group (RTOG) recursive partitioning prognostic subgroups, which includes patient age, KPS, extent of resection and neurological function.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age greater than or equal to 18 years.

Histologically confirmed supratentorial Glioblastoma multiforme.

Karnofsky performance >60.

Patient must be a candidate for radiotherapy.

Ability of subject or Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

Patients with other cancers excluding non-melanomatous skin cancers or carcinoma in situ.

Gliadel wafer placement at the time of surgery.

Pregnancy because radiation has the potential for teratogenic or abortifacient effects.

<TAB><TAB>

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving radiation therapy for Glioblastoma multiforme (GBM). Primary clinical.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2004-06-22 (Actual)

PRIMARY OUTCOMES:
To determine if an increase in urinary VEGF and MMP level, from the end of treatment to a patient's one-month follow-up examination following radiotherapy is predictive of one-year recurrence in patients with Glioblastoma multiforme | one year
  Determine the whether VEGF and MMP level measurements aid in predicting tumor recurrence at 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin A Camphausen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2004-C-0200.html